CLINICAL TRIAL: NCT04284748
Title: Effect of Plyometric Training With Blood Flow Restriction on Muscle Strength and Function After Anterior Cruciate Ligament Reconstruction
Brief Title: Effect of Blood Flow Restriction Training on Patient With Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERDAR DEMIRCI, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-180096
Record Dates: First submitted 2020-01-07; First posted 2020-02-26 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2018-11

CONDITIONS: Anterior Cruciate Ligament Injuries; Atrophy; Muscle Weakness
Keywords: anterior cruciate ligament reconstruction; atrophy; knee function
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Atrophy; Muscle Weakness | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric training with blood flow restriction (Experimental): Routine physiotherapy program + Plyometric training with blood flow restriction, 3 days a week for 8 weeks Jump in functional squat system (30+15+15+15= 75 rep) Lunge jump (30 rep) Side jump (30 rep) Box jump (15 rep) Exercises to be added after 4 weeks; Square jump (15 rep) One leg hop (15 rep)
  Interventions: Other: Plyometric exercise with blood flow restriction; Other: Routine physiotherapy program
- Plyometric training (Active Comparator): Routine physiotherapy program + Plyometric training 3 days a week for 8 weeks Jump in functional squat system (30+15+15+15= 75 rep) Lunge jump (30 rep) Side jump (30 rep) Box jump (15 rep) Exercises to be added after 4 weeks; Square jump (15 rep) One leg hop (15 rep)
  Interventions: Other: Plyometric exercise; Other: Routine physiotherapy program

INTERVENTIONS:
Other: Plyometric exercise with blood flow restriction — Blood flow restriction training is an exercise protocol based on the method of limiting blood flow with external pressure by pneumatic tourniquet from the proximal of the muscle to be strengthened. Blood flow restriction (Occlusion) during pliometric exercises for 8 weeks, a pneumatic tourniquet (Kaatsu Master) proximal to the thigh will be applied to each patient within a safe pressure range. The pressure to be applied to the patient will be calculated with the following formula described in the literature.
  Pressure = 0.5 x (systolic blood pressure) + 2 x (thigh circumference) + 5 Application will be done for a maximum of 15 minutes, then rest for 10-15 minutes and other exercises will continue.
  Plyometric training with blood flow restriction. Jump in functional squat system (30+15+15+15= 75 rep) Lunge jump (30 rep) Side jump (30 rep) Box jump (15 rep) Exercises to be added after 4 weeks; Square jump (15 rep) One leg hop (15 rep)
  Arms: Plyometric training with blood flow restriction
Other: Plyometric exercise — Plyometric training Jump in functional squat system (30+15+15+15= 75 rep) Lunge jump (30 rep) Side jump (30 rep) Box jump (15 rep) Exercises to be added after 4 weeks; Square jump (15 rep) One leg hop (15 rep)
  Arms: Plyometric training
Other: Routine physiotherapy program — Anterior and lateral plan exercise (3x10 rep) Open kinetic quadriceps and hamstring strengthening exercise (3x10 rep) Lunge exercises on different ground (3x10 rep) Single leg squat exercise on different ground (3x10 rep) Anterior and lateral walking exercise in a squatting position with an exercise band (40 step) Balance and proprioceptive exercises

SUMMARY:
This study investigates the effects of plyometric training with blood flow restriction on muscular strength, quadriceps thickness and knee joint function in patients with muscle weakness and atrophy (quadriceps muscle and hamstring muscle) after anterior cruciate ligament reconstruction. Persons who completed a 12-week routine rehabilitation program after anterior cruciate ligament reconstruction will be included in the study. In the study group, plyometric exercises will be performed with blood flow restriction in the operated side for 8 weeks. In the control group, the same plyometric exercises will be performed without any application.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) rupture is one of the most common sports injuries. Surgical procedure is usually performed after injury. After ACL surgery, patients experience problems such as pain, impaired knee function, and especially quadriceps muscle weakness and atrophy. Quadriceps atrophy has been shown to persist for years despite rehabilitation programs. Therefore, rehabilitation programs after ACL reconstruction play an important role in ensuring return to sports and reducing postoperative complications. In general, ACL rehabilitation can be divided into early and late periods. In the early period, while focusing on the solution of the primary problems related to the knee (pain, edema, joint movement limitation, quadriceps muscle weakness, and antalgic gait), the focus is on the patient's preparation for returning to sports activities. Running, jumping and agility training are the exercise approaches of late phase rehabilitation. These exercises include pliometric activities that trigger the stretch-shortening cycle of the lower extremity extensor muscles. Pliometric exercises after anterior cruciate ligament reconstruction may improve lower extremity muscle strength and knee function and increase the rate of return to sports, but there is not enough study in this area. Under normal conditions, 6-12 repetitive weight-lifting exercises at a density of at least 65% of a maximum repetition are recommended to increase strength in a muscle and achieve hypertrophy. However, it takes approximately 4-6 months for the ligament to mature and bear weight after surgery. For this reason, high intensity strengthening training is not used in the early period of rehabilitation to protect the graft that is recovering after surgery and the training is started from low intensity and increased gradually. Recent studies suggest that muscle hypertrophy occurs with low-intensity exercises (20-30% of a maximum repetition) with blood flow restriction, also known as KAATSU training or occlusion training. Because blood flow restriction training allows the benefits of high intensity training to be obtained at a much lower intensity. In the literature, the effectiveness of many different exercise programs after ACL reconstruction was investigated. However, no study investigating the effect of blood flow restriction plyometric exercise training on ACL rehabilitation on muscle strength and function was found. This study will be conducted to investigate the contribution of low-density plyometric training with blood flow restriction to atrophy, muscle strength, function and return to sports.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 year
* Volunteering to participate in the study
* Patients who had unilateral anterior cruciate ligament surgery with hamstring tendon auto graft and completed 12 weeks of rehabilitation program

Exclusion Criteria:

* Systemic or neurological problems
* Endothelial dysfunction
* Peripheral vascular diseases and history of deep vein thrombosis
* Active infection, cancer, pregnant,
* Posterior cruciate ligament tear, medial or lateral collateral ligament tear and knee cartilage damage

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle thickness and rectus femoris cross-sectional ares | 8 week
  Thickness of rectus femoris, vastus medialis obliques, vastus lateralis muscles and cross-sectional area of rectus femoris were measured using a B-mode ultrasound device with a 9L4 linear probe before and after plyometric training.
Hamstring and quadriceps muscle strength | 8 week
  Quadriceps and hamstring muscle strength (isometric, concentric and eccentric) were evaluated with an isokinetic dynamometer (IsoMed2000 D&R GmbH, Germany) before and plyometric training.

SECONDARY OUTCOMES:
Vertical jump test (VJT) | 8 week
  The assessment leg was positioned closest to the wall. The point where the patient reached out with his hand in elbow extension was marked. Then, the patients were standing on assessment foot, one foot length away from the wall. They jumped vertically and made a mark on the wall with a marker. The distance between the patient's jump and touch point and the starting point was measured with tape. This test was performed three times for each leg, and the average of the three values was calculated. The VJT uses the limb symmetry index for VJT calculated as ([reconstructed limb-hop distance/ contralateral limb-hop distance] x 100).
One leg hop test (OLHT) | 8 week
  Participants stood on one leg with toes behind a mark on the floor and performed one hop as far as possible along a straight line, landing on the same foot. The test started with the uninvolved limb followed by the involved limb. The distance in centimeter was measured. This test was performed three times for each leg, and the average of the three values was calculated. The OLHT uses the limb symmetry index for OLHT calculated as ([reconstructed limb-hop distance/ contralateral limb-hop distance] x 100).
Single leg triple hop test (SLTHT) | 8 week
  Participants stood on one leg with toes behind a mark on the floor and performed triple hop as far as possible along a straight line, landing on the same foot. The test started with the uninvolved limb followed by the involved limb. The distance in centimeter was measured. This test was performed three times for each leg, and the average of the three values was calculated. The SLTHT uses the limb symmetry index for SLTHT calculated as ([reconstructed limb-hop distance/ contralateral limb-hop distance] x 100).
Y balance test | 8 week
  The dynamic balances of the individuals were evaluated with the Y balance test (Modified Star Excursion Balance Test, SEBT). The test was carried out with a Y balance test kit consisting of three pipes marked with a distance in cm, with the front pipe and other pipes 135 ° and the pipes 90 ° from the back. Before the evaluation, the test was shown to the participant once and they were given a chance to try in all 3 directions. The test started with the uninvolved leg followed by the involved leg. The test was repeated 3 times in all directions and the mean was recorded. The average scores were divided by the leg length of the individual (the distance between the sipina iliaca anterior superior and the medial malleol), multiplied by 100 and recorded to normalize the reach distances in all directions.
Knee Documentation Committee (IKDC) Questionnaire | 8 week
  IKDC, a valid and reliable measure for ACL injury and ACLR (ICC = 0.91), contains ten items related to knee symptoms in addition to daily and sports activities. Scores range from 0 to 100 with higher scores indicating less disability.
Knee Injury and Osteoarthritis Outcome Questionnaire (KOOS) | 8 week
  The Turkish version of the KOOS scale (ICC> 0.75), a valid reliable measurement, was used to evaluate pain, functional status, daily life activity and quality of life. The scale has 5 subtitles: pain, daily life activities, sports and leisure activities, functional status and string-related quality of life. Each subtest is scored between 0 and 100. The higher score indicates better knee function.
Tampa Kinesiophobia Scale | 8 week
  The Turkish validity and reliability study Tampa Kinesiophobia Scale was used to evaluate individuals' fear and avoidance of movement. The test is calculated by 17-point Likert scoring. The individual scores between 17-68 and as the score increases, the level of kinesiophobia increases.
Anterior Cruciate Ligament Return to Sport After Injury Scale (ACL-RSI) | 8 week
  The Turkish version of the ACL-RSI scale was used to evaluate individuals' return to sports rate. The scale consisting of 12 questions, scored between 0-10 according to the visual analog scale; emotions consist of performance self-confidence and risk assessment subtitles. High scores show the subjective perception of individuals about returning to sports

CONTACTS AND LOCATIONS:
Overall Officials: Egemen Turhan, MD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Department of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available